CLINICAL TRIAL: NCT06689618
Title: Effects of Whole-body Electrical Muscle Stimulation Exercise on Spinal Motoneuronal Activation in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kristina Kelly, Assistant Research Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2116666
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Aging; Sarcopenia; Sarcopenia in Elderly
Keywords: Aging; Motoneuronal Activation; Electrical Stimulation; Whole-Body Stimulation; Sarcopenia; Exercise Intervention; Exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Enrolled participants will undergo pre-test assessments within 2-4 days before and after the intervention period. The pre-test assessment visit will be scheduled for 3.5 hours, and the post-test assessment visit for 2.5 hours, reflecting that the pre-test visit will incorporate consenting and screening procedures. The intervention will consist of 2 visits per week for 4 weeks; each intervention visit will be scheduled for 1.5 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy Adults (Experimental): All participants will receive the WB-EMS Exercise intervention 2 times per week for 4 weeks. Participants will only perform leveled exercise programs in the "Strength" Training Mode. These programs are 20-minute videos led by exercise professionals. They are full-body workouts with no one muscle group receiving more attention than another. They consist of 10-12 exercises performed for 14 repetitions. Each repetition takes 4 seconds to complete (the time that the stimulation is "on") and is followed by a 4 second rest (the time that the stimulation is "off"). All exercises occur in a double-limb stance position. Most exercises occur with feet in wide base of support, hips width or more apart. All exercises are modifiable by the healthcare professional administering and monitoring the intervention based on participant's safe and available range of motion (i.e. arm movements, torso positions, extent of knee bend).
  Interventions: Device: Exercise

INTERVENTIONS:
Device: Exercise — The WB-EMS Device is a fitness device that delivers whole-body electrical muscle stimulation in conjunction with exercise programs. After donning a base layer consisting of fitted shorts and shirt, a vest, shorts, and arm straps with integrated electrodes mapped to major muscle groups (biceps, triceps, pectorals, abdominals, periscapular musculature, paraspinal musculature, gluteus musculature, quadriceps, and hamstrings) are donned. The suit connects to an impulse pack that communicates with the Katalyst iPad App to deliver the programmed stimulation to the participant. Within the Katalyst App, there are leveled exercise programs where low levels (i.e. Level 1 and 2) are simple movements and higher levels (i.e. Levels 3, 4, and 5) have more complex and dynamic movements. There is complete user control of the stimulation level of each individual muscle group to tailor to participant responses and tolerance.
  Other Names: Whole-Body Electrical Stimulation

SUMMARY:
During this pilot study, the investigators will examine the effects of whole-body electrical muscle stimulation exercise (WB-EMS Exercise) on motoneuronal activation in healthy adults, which typically decreases with age. The investigators will also test whether WB-EMS Exercise will improve measures of physical function. Participants will undergo clinical and electrophysiologic testing before and after the WB-EMS Exercise intervention. The WB-EMS Exercise intervention will be delivered two times per week for four weeks. The hypothesis is that whole-body electrical muscle stimulation combined with physical exercise (WB-EMS Exercise) could bypass the problem of insufficient motoneuronal activation to improve exercise effect in older adults.

DETAILED DESCRIPTION:
During this pilot study, the investigators will examine the effects of whole-body electrical muscle stimulation exercise (WB-EMS Exercise) on motoneuronal activation in healthy adults, which typically decreases with age. The investigators will also test whether WB-EMS Exercise will improve measures of physical function. The intervention consists of WB-EMS Exercise twice a week for four weeks. The investigators will use decomposition electromyography, interpolated twitch technique, and clinical measures to assess pre- and post-treatment motoneuronal activation and physical functioning. Correlation matrices will be performed associating the measures of motoneuronal activation to the measures of physical function (pre-intervention values, post-intervention values, and change values). At the conclusion of the study, expected outcomes include that whole-body electrical muscle stimulation combined with physical exercise (WB-EMS Exercise) could bypass the problem of insufficient motoneuronal activation to improve exercise effect in older adults. This project represents early work to uncover motoneuronal mechanisms of WB-EMS Exercise in older adults. An intervention that combines voluntary and involuntary activation of motoneurons to enhance the effectiveness of exercise could have significant impact in maximizing the functional independence of an aging population.

ELIGIBILITY:
Inclusion Criteria:

* Age (65 years or older) for healthy older adults and between 18-39 for healthy younger adults
* Ambulatory without an assistive device
* More than anti-gravity strength in major muscle groups as assessed by manual muscle testing
* Medical clearance to participate in an exercise program
* Ability to conform to the requirements of the study (i.e. attendance at assessment and intervention visits, maintain current level of non-study physical activity for the duration of the study, no intention to relocate mid-study)

Exclusion Criteria:

* Regular use of an assistive device for mobility (i.e. cane, walker, wheelchair)
* Presence of a pacemaker, metal implants, or other implanted medical devices that could impact participant safety during WB-EMS intervention
* Known pregnancy at the time of screening
* Presence of unstable acute or chronic disease (i.e. renal failure, rheumatologic disease cardia arrhythmia, neoplasm, uncontrolled hypertension)
* Presence of terminal disease (i.e. receiving hospice services)
* Current of previous use of any drugs known to influence muscle mass or performance within 6 months; these may include but are not limited to anabolic steroids, IGF01, growth hormone, replacement and androgen therapy, anti-androgen therapy.
* Known neuromuscular or neurologic condition affecting somatosensory or motor function/control (i.e. motor neuron disease, muscle disease, severe peripheral neuropathy, NMJ disease, Parkinson's disease, Multiple Sclerosis, h/o stroke, TBI, SCI, ataxia, apraxia, hemiplegia, etc.)
* Musculoskeletal condition or surgery in the past year that would confound results of exercise interventions (i.e. TKA, THA, RTC repair, spinal fusion)
* Other medical conditions, signs, or symptoms that would interfere with study conduct or interpretation of results as determined by a PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in motor unit firing rates of the vastus lateralis using decomposition electromyography (dEMG) | Measured within 3 days of starting the intervention and within 3 days of completing the intervention
  Decomposition electromyography (dEMG) is a measurement of motor unit activity; a surface electrode will be placed over the vastus lateralis in the thigh and participants will be asked to activate that muscle.
Mean change from baseline in central activation ratio of the vastus lateralis using interpolated twitch technique (ITT) | Measured within 3 days of starting the intervention and within 3 days of completing the intervention
  The central activation ratio (CAR) is a representation of how completely a person can voluntarily access their maximum force production capacity. Surface electrodes will be placed over the vastus lateralis in the thigh and participants will be asked to activate that muscle.

SECONDARY OUTCOMES:
Mean change from baseline in mobility testing | Measured within 3 days of starting the intervention and within 3 days of completing the intervention
  To capture changes in common functional movements relevant to maintenance of independence for older adults, the investigators will collect data on gait speed (10-m walk/run test), stair negotiation (4-stair ascent and descent), rising from/lowering to a chair (30 second sit to stand), and lowering to/rising from the floor (floor transfer test).
Mean change from baseline in balance testing | Measured within 3 days of starting the intervention and within 3 days of completing the intervention
  The Balance Outcome Measure for Elder Rehabilitation (BOOMER) is an older adult-specific measure of balance. It is a composite test consisting of a Step Test (tapping a step with one foot as many times as safely possible in 15 seconds), the Timed Up and Go (TUG; rise from a chair, walk 3 meters, turn around, and return to sitting in chair), the Functional Reach Test (FRT; standing forward reach with arms outstretched as far as a person can control), and a Timed Static Stance (narrow stance, eyes closed for up to 90 seconds). Participants will also complete the Single Leg Hop test and the Star Excursion Test.
Treatment Feedback Questionnaire | Measured within 3 days of completing the intervention
  The Treatment Feedback Questionnaire was created by the principal investigator to systematically collect meaningful feedback from the participants regarding their opinions, impressions, and recommendations about the WB-EMS Exercise intervention. This is part of an ongoing effort to develop exercise interventions that are effective and patient-centered and can be adopted and sustained to promote long-term health.

CONTACTS AND LOCATIONS:
Locations (1):
- NextGen Precision Health Building, Clinical and Translational Science Unit, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No